CLINICAL TRIAL: NCT05672680
Title: Transabdominal Plane (TAP) Blocks for Inguinal Hernia Repairs
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Celia M. Divino, The Edelman Professor of Surgery, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY-19-00677
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Normal Saline:
  For patients weighing <100 kg, a total of 50 ml ((25 ml on each side of the abdominal wall) will be received. If patients weigh>100 kg, a total of 60 ml (30ml on each side of the abdominal wall) will be received.
  Interventions: Drug: Placebo; Procedure: TAP block
- Experimental (Experimental): 0.25% bupivacaine: For patients weighing <100 kg, a total of 50 ml ((25 ml on each side of the abdominal wall) will be received. If patients weigh>100 kg, a total of 60 ml (30ml on each side of the abdominal wall) will be received.
  Interventions: Drug: 0.25% Bupivacaine; Procedure: TAP block

INTERVENTIONS:
Drug: 0.25% Bupivacaine — received during TAP block
  Arms: Experimental
Drug: Placebo — placebo equivalent
  Arms: Placebo
Procedure: TAP block — The intervention is a transabdominal plane (TAP) block given in the abdomen to block pain receptors on nerves -during surgery can presumably decrease postoperative pain. Currently, TAP blocks are approved for use and performed based on surgeon preference (e.g. some surgeons perform them on every case, others variably, etc.).

SUMMARY:
The aim of this double-blind clinical trial is to examine outcomes and pain control after surgery in patients who underwent laparoscopic inguinal hernia repair (IHR) with the use of perioperative transabdominal plane (TAP) block.

Research Question: Does transabdominal plane block improve pain when undergoing inguinal hernia repair? The endpoints include whether preoperative TAP blocks improve pain score (primary end point) and decrease opioid use (secondary endpoint) after an inguinal hernia repair. Other end points- complications after surgery.

DETAILED DESCRIPTION:
Protocol:

After receiving approval for the study, the researchers will conduct a prospective single institution randomized clinical trial assessing if using a TAP block perioperatively can reduce pain scores after surgery. Other endpoints include whether there are differences in pain medication usage and complications.

Patients will be screened by research team members and attending surgeons. If the patient is interested, the researchers will consent the participants for the study after understanding the study details, procedures, and expectations. The researchers will then consent using IRB approved study consent forms and procedures. Patients will undergo a laparoscopic inguinal hernia repair according to standard procedures. The study will assess if a TAP block impacts pain scores. Patients will be randomized to receive the intervention or placebo. Sequentially numbered sealed opaque envelopes with group allocation inside will alert the anesthesiologist & surgeon to order Tap block composed of 0.25% bupivacaine or placebo (normal saline).

Inguinal hernia repair will be performed in standard fashion that each individual surgeon is familiar with. No additional tests or blood work outside the standard of care for IHR will be performed for research purposes. In addition, some patients will be given TAP blocks before surgery to help in pain management. Patients will be discharged with a worksheet on which the participants are to record analgesic use and pain scores on postoperative days one, two, three and four. The participants are expected to bring the completed log to their two-week follow up visit with their surgeon. Patients may also expect to receive a phone call from a member of the surgical team to remind them to record these metrics.

The TAP block is done pre-procedure using 0.25% bupivacaine. If patients weigh<100 kg, the patients will receive a total of 50 ml (25 ml on each side of the abdominal wall). If patients weigh>100 kg, the patients will receive a total of 60 ml (30ml on each side of the abdominal wall). The TAP plane is identified using ultrasound. All anesthesiologists (not surgeons) working with the attendings involved in this study have been trained in this technique; it is a routine part of their practice. It is anesthesiologists who will be performing the block.

Patients will be discharged with a worksheet /survey on which the patients are to record analgesic use and pain scores on postoperative days one, two, three and four. The patients are expected to bring the completed log to their two-week follow up visit.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing laparoscopic inguinal hernia repair at the Mount Sinai Hospital

Exclusion Criteria:

* patients who are younger than 18 years old,
* have a history of chronic opiate usage, liver or kidney disease, pain syndromes,
* allergy to bupivacaine,
* are pregnant or
* are unable to independently give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Celia M Divino, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Data will be published in aggregate form without any PHI or references to the patient so as to keep identifying information secure.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment performed in outpatient office from 12/9/2019 to 07/23/2023.
Groups:
- Placebo: Normal Saline:
  For patients weighing <100 kg, a total of 50 ml ((25 ml on each side of the abdominal wall) will be received. If patients weigh>100 kg, a total of 60 ml (30ml on each side of the abdominal wall) will be received.
  Placebo: placebo equivalent
  TAP block: The intervention is a transabdominal plane (TAP) block given in the abdomen to block pain receptors on nerves -during surgery can presumably decrease postoperative pain. Currently, TAP blocks are approved for use and performed based on surgeon preference (e.g. some surgeons perform them on every case, others variably, etc.).
Period: Overall Study
Arm/Group | Placebo | Experimental
Started | 50 | 50
Completed | 44 | 46
Not Completed | 6 | 4
Not completed — Patient Did Not Complete the Form | 5 | 4
Not completed — Procedure Aborted | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Experimental | Total
Number analyzed (Participants) | 44 | 46 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.07 (13.67) | 56.42 (15.78) | 57.24 (14.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 41 | 44 | 85
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Pain Score at Rest
Description: On the pain score instrument, patients will score their pain score at rest. The full scale is scored between 1-10, with higher score indicating more pain.
Time Frame: on post-op days 1, 2, 3, and 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 44 | 46
score on a scale
  post-op day 1 | 4.31 (2.46) | 4.55 (2.70)
  post-op day 2 | 4.21 (2.49) | 4.53 (2.61)
  post-op day 3 | 3.53 (2.39) | 3.77 (2.49)
  post-op day 4 | 2.92 (2.39) | 3.19 (2.46)

2. Primary Outcome: Pain Score at Rest
Description: as for outcome 1
Time Frame: All post-op (average 4 days)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 44 | 46
score on a scale | 3.75 (2.48) | 4.01 (2.65)

3. Primary Outcome: Pain Score at Movement
Description: On the pain score instrument, patients will score their pain score at movement. The full scale is scored between 1-10, with higher score indicating more pain.
Time Frame: on post-op days 1, 2, 3, and 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 44 | 46
score on a scale
  post-op day 1 | 5.84 (2.42) | 6.35 (2.54)
  post-op day 2 | 5.47 (2.56) | 6.16 (2.55)
  post-op day 3 | 4.65 (2.21) | 4.99 (2.51)
  post-op day 4 | 3.71 (2.37) | 4.31 (2.53)

4. Primary Outcome: Pain Score at Movement
Description: as for outcome 3
Time Frame: All post-op (average 4 days)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 44 | 46
score on a scale | 4.93 (2.51) | 5.46 (2.67)

5. Secondary Outcome: Number of Opioid Pills
Description: Patients recorded the number of opioid pills taken.
Time Frame: on post-op days 1, 2, 3, and 4
Measure: Mean (Standard Deviation); unit: number of pills
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 44 | 46
number of pills
  post-op day 1 | 1.29 (1.47) | 1.52 (1.28)
  post-op day 2 | 1.25 (1.62) | 1.35 (1.48)
  post-op day 3 | 0.88 (1.45) | 0.60 (1.10)
  post-op day 4 | 1.21 (1.54) | 0.77 (1.26)

6. Secondary Outcome: Number of Opioid Pills
Description: Patients recorded the number of opioid pills taken.
Time Frame: All post-op (average 4 days)
Measure: Mean (Standard Deviation); unit: number of pills
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 44 | 46
number of pills | 1.16 (1.52) | 1.06 (1.33)

7. Secondary Outcome: Number of Non-opioid Pain Medication
Description: Patients recorded the number of non-opioid pills taken for pain control.
Time Frame: on post-op days 1, 2, 3, and 4
Measure: Mean (Standard Deviation); unit: number of pills
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 44 | 46
number of pills
  post-op day 1 | 0.76 (1.03) | 0.71 (1.09)
  post-op day 2 | 1.07 (1.22) | 0.78 (1.05)
  post-op day 3 | 0.85 (1.04) | 0.77 (0.96)
  post-op day 4 | 0.77 (0.98) | 0.65 (0.82)

8. Secondary Outcome: Number of Non-opioid Pain Medication
Description: Patients recorded the number of non-opioid pills taken for pain control.
Time Frame: All post-op (average 4 days)
Measure: Mean (Standard Deviation); unit: number of pills
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 44 | 46
number of pills | 0.86 (1.07) | 0.73 (0.98)

9. Secondary Outcome: Number of Intraoperative Complications
Description: Chart review complications recorded. These are considered expected intraoperative complications and are not considered as adverse events based on research procedures.
Time Frame: up to 2 weeks post-surgery
Measure: Number; unit: number of complications
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 44 | 46
number of complications
  Mortality | 0 | 0
  Urinary Retention | 1 | 2
  Early Recurrence | 0 | 1
  Hematoma | 0 | 1
  Induration | 1 | 1

10. Secondary Outcome: Number of Participants With Contents in the Hernia
Description: Number of participants with contents in the hernia, specifically bowel, lipoma, omentum, and bladder.
Time Frame: during procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 44 | 46
Participants
  None | 33 | 39
  Bowel | 1 | 0
  Lipoma | 10 | 6
  Omentum | 0 | 1
  Bladder | 0 | 0

11. Secondary Outcome: Number of Surgical Tacks Used Per Repair
Description: Number of tacks used in bilateral hernia surgery per repair. The more tacks used can be associated with increased pain.
Time Frame: during procedure
Population: There were a number of participants that were missing this data. This is due to human error for not inputting the information.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 44 | 46
Participants
  4 | 16 | 12
  5 | 0 | 3
  6 | 18 | 15
  Data not collected | 10 | 16

12. Secondary Outcome: Procedure Time
Description: Procedure duration in minutes.
Time Frame: during procedure
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 44 | 46
Minutes | 72.7 (19.13) | 78.54 (27.20)

13. Secondary Outcome: Number of Participants With Greater or Less Than 25 Milliliters Estimated Blood Loss
Description: Number of participants with greater or less than 25 milliliters estimated blood loss recorded during procedure.
Time Frame: during procedure
Population: A participant was missing this data. This is due to human error for not inputting the information.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 44 | 46
Participants
  Less than 25 milliliters | 38 | 39
  Greater than or equal to 25 milliliters | 5 | 7
  Data not collected | 1 | 0

14. Secondary Outcome: Number of Patients Per Anesthesiologist
Description: The number of patients handled per anesthesiologist.
Time Frame: during procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 44 | 46
Participants
  Anesthesiologist 1 | 18 | 21
  Anesthesiologist 2 | 3 | 2
  Anesthesiologist 3 | 7 | 4
  Anesthesiologist 4 | 16 | 19

ADVERSE EVENTS:
Time Frame: up to 2 weeks post-surgery
Arm/Group | Placebo | Experimental
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/46
Other Adverse Events (participants affected / at risk) | 0/44 | 0/46

LIMITATIONS AND CAVEATS:
Demographic information, like race and ethnicity was not obtained.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT05672680/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-29): https://cdn.clinicaltrials.gov/large-docs/80/NCT05672680/ICF_001.pdf